CLINICAL TRIAL: NCT06053931
Title: The Effect of Music on Neonatal Stress, Mother's Breastfeeding Success and Comfort During Breastfeeding: a Randomized Controlled Trial
Brief Title: The Effect of Music on Neonatal Stress, Mother's Breastfeeding Success and Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Manisa Celal Bayar University
Record Dates: First submitted 2023-09-10; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Music; Breastfeeding; Newborn; Mother
Keywords: White noise; Lullaby; neonatal stress; comfort
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A total of 90 mothers and newborns, 30 lullaby, 30 white noise and 30 control groups, will constituted the sample of the study
Who Masked: Participant
Masking Description: The population of the research is consisted of mothers who have just given birth and are hospitalized in the obstetrics and gynecology service at Izmir Bakırçay University Çiğli Training and Research Hospital.
  No sample selection is made in the research, and all mothers who meet the inclusion criteria and accept the research is constituted the sample.
  Randomization will be provided to newborns and mothers using the simple randomization method according to their protocol numbers and by using the website https://www.randomizer.org/.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The women will fill out an descriptive characteristics questionnaire, which include questions such as age, education and employment status, number of pregnancies and children etc. Mothers will be asked to mark before breastfeeding on their comfort on the Visual Analog Scale. The number "0" on the scale indicates that it is not comfortable at all, and the number "10" indicates that the comfort is complete.The baby's stress level will measure with the "Newborn Stress Scale" before breastfeeding. While the mother is breastfeeding her baby, the breastfeeding process will be evaluated by the researcher with the "LATCH Breastfeeding Assessment Tool". Baby's stress level will be evaluated at the 1st minute of breastfeeding with the "Newborn Stress Scale". After the breastfeeding process is completed, the mother will be asked to fill out the "Visual Analog Scale" again to evaluate her comfort.
- Lullaby group (Experimental): The women will fill out an descriptive characteristics questionnaire. Mothers will be asked to mark before breastfeeding on their comfort on the scale.
  The baby's stress level will measure with the "Newborn Stress Scale" before breastfeeding.
  Before the mother starts breastfeeding her baby, lullaby music will be turned on to help the baby relax during 2 minutes.
  During the breastfeeding process, music will be played to the baby and mother for approximately 15 minutes.
  The baby will be observed by the researcher at the first minute of breastfeeding, and the Newborn Stress Scale will be filled in again.
  The LATCH assessment will be done within the first 15 minutes of breastfeeding. After breastfeeding is over, they will be asked to fill in the "Visual Analog Scale" in order to evaluate the comfort of the mother.
  Interventions: Behavioral: lullaby music
- White noise group (Experimental): The women will fill out an descriptive characteristics questionnaire. Mothers will be asked to mark before breastfeeding on their comfort on the scale.
  The baby's stress level will measure with the "Newborn Stress Scale" before breastfeeding.
  Before the mother starts breastfeeding her baby, white noise music will be turned on to help the baby relax during 2 minutes During the breastfeeding process, music will be played to the baby and mother for approximately 15 minutes.
  The baby will be observed by the researcher at the first minute of breastfeeding, and the Newborn Stress Scale will be filled in again.
  The LATCH assessment will be done within the first 15 minutes of breastfeeding. After breastfeeding is over, they will be asked to fill in the "Visual Analog Scale" in order to evaluate the comfort of the mother.
  Interventions: Behavioral: white noise music

INTERVENTIONS:
Behavioral: white noise music — Before the mother starts breastfeeding her baby, white noise music will be turned on to help the baby relax during 2 minutes and during the breastfeeding process, music will be played to the baby and mother for approximately 15 minutes.
  (https://www.youtube.com/watch?v=5NFHiKMCPvw&t=6478s).
  Other Names: white noise
  Arms: White noise group
Behavioral: lullaby music — Before the mother starts breastfeeding her baby, lullaby music will be turned on to help the baby relax during 2 minutes and during the breastfeeding process, music will be played to the baby and mother for approximately 15 minutes.
  (https://www.youtube.com/watch?v=h0QO8bgysPg)
  Other Names: lullaby
  Arms: Lullaby group

SUMMARY:
In the literature, music plays an energizing, soothing, stimulating and awakening role for the newborn, and at the same time, music has the potential to wake up a lethargic and withdrawn baby and calm a crying, restless baby. In addition, it is stated that relaxing music in the early postpartum period supports breastfeeding behaviors of mother and baby. It is stated that lullabies positively affect the newborn's relaxation, falling asleep, and mother-baby communication. however, it facilitates sleep due to its monotonous, emotional and repetitive melody structure, slow tempo and relaxing effect. The sound called white noise is a humming, monotonous and constantly used sound that suppresses the disturbing sounds coming from the environment and has a calming feature. In the literature, it has been found that white noise played to infants with colic reduces crying.

The aim of this study is to determine the effects of lullabies and white noise music played during breastfeeding of the newborn on newborn stress, breastfeeding success and mother's comfort. This study was planned as a randomized controlled trial with term newborns 24 hours after birth.

DETAILED DESCRIPTION:
The hypotheses are presented below;

H1- White noise music played during breastfeeding reduces newborn stress compared to the control group.

H2- White noise music played during breastfeeding increases breastfeeding success compared to the control group.

H3- White noise music played during breastfeeding increases comfort of the mother compared to the control group.

H4- Lullaby music played during breastfeeding reduces newborn stress compared to the control group.

H5- Lullaby music played during breastfeeding increases breastfeeding success compared to the control group.

H6- Lullaby music played during breastfeeding increases comfort of the mother compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Able to speak Turkish,
* Breastfeeding mothers
* Term and healthy newborn (born at 38-42 weeks, weighing 2500-4000 g, born with an APGAR of 7 or more, without any known congenital disease)

Exclusion Criteria:

* mothers who do not agree to participate in the research
* mother has a condition that prevents breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
newborn stress level in white noise group | from pre-intervention to 2 minutes after listening to white noise music.
  Change in newborn stress level from pre-intervention to 2 minutes after listening to white noise music in the first minute of breastfeeding. "Newborn Stress Scale" including facial expression, color, respiration, activity level, consolation, muscle tone, extremities, and posture. Each parameter was scored on a scale of 0-2. The minimum score was 0, and the maximum score was 16 for this scale, where a higher score represented increased stress levels in newborn.
newborn stress level in lullaby group | from pre-intervention to 2 minutes after listening to lullaby.
  Change in newborn stress level from pre-intervention to 2 minutes after listening to lullaby.
  "Newborn Stress Scale" including facial expression, color, respiration, activity level, consolation, muscle tone, extremities, and posture. Each parameter was scored on a scale of 0-2. The minimum score was 0, and the maximum score was 16 for this scale, where a higher score represented increased stress levels in newborn.
mother's comfort in white noise group | from pre-intervention to 15 minutes after listening to white noise music
  Change in mother's comfort from pre-intervention to 15 minutes after listening to white noise music during breastfeeding. The number "0" on the the Visual Analog Scale indicates that it is not comfortable at all, the comfort increases as the numbers get larger, and the number "10" indicates that the comfort is complete.
mother's comfort in lullaby group | from pre-intervention to 15 minutes after listening to lullaby.
  Change in mother's comfort from pre-intervention to 15 minutes after listening to lullaby during breastfeeding.

SECONDARY OUTCOMES:
breastfeeding success in white noise group | At the 15th minute of breastfeeding
  At the 15th minute of breastfeeding in white noise group, breastfeeding success will be evaluated using the LATCH Breastfeeding Assessment Tool.
  LATCH is a breastfeeding charting system that provides a systematic method for gathering information about individual breastfeeding sessions. The system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding. Each letter of the acronym LATCH denotes an area of assessment. "L" is for how well the infant latches onto the breast. "A" is for the amount of audible swallowing noted. "T" is for the mother's nipple type. "C" is for the mother's level of comfort. "H" is for the amount of help the mother needs to hold her infant to the breast.
breastfeeding success in lullaby group | At the 15th minute of breastfeeding
  At the 15th minute of breastfeeding in lullaby group, breastfeeding success will be evaluated using the LATCH Breastfeeding Assessment Tool.
  LATCH is a breastfeeding charting system that provides a systematic method for gathering information about individual breastfeeding sessions. The system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding. Each letter of the acronym LATCH denotes an area of assessment. "L" is for how well the infant latches onto the breast. "A" is for the amount of audible swallowing noted. "T" is for the mother's nipple type. "C" is for the mother's level of comfort. "H" is for the amount of help the mother needs to hold her infant to the breast.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı KARAKUŞ SELÇUK, PhD, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No